CLINICAL TRIAL: NCT04609228
Title: Cardiac Surgery Outcomes in Blood-transfusion Acceptors and no Acceptors: a Retrospective Cohort Study
Brief Title: Cardiac Surgery Outcomes in Blood-transfusion Acceptors and no Acceptors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-TRA-2020-36
Record Dates: First submitted 2020-10-15; First posted 2020-10-30 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Thoracic Surgery; Blood Transfusion; Hemoglobinemia; Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blood-transfusion non-acceptors: Blood-transfusion non-acceptors
  Interventions: Other: Non-acceptance of blood-transfusions
- Blood-transfusion acceptors: Blood-transfusion acceptors
  Interventions: Other: Acceptance of blood-transfusions

INTERVENTIONS:
Other: Non-acceptance of blood-transfusions — Patients who do not accept blood products transfusions
  Groups: Blood-transfusion non-acceptors
Other: Acceptance of blood-transfusions — Patients who accept blood products transfusions
  Groups: Blood-transfusion acceptors

SUMMARY:
The primary objective of this study is to analyze mortality after cardiac surgery in blood-transfusion non-acceptors (BTNA), and the secondary one to perform an adjusted comparison with a blood-transfusion acceptors (BTA) matched cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing heart surgery in our hospital from 2009 to June 2020

Exclusion Criteria:

* Preoperative hemoglobin lower than 120g/L
* EuroSCORE-II higher than 20%
* Heart transplant
* Assist device implantation
* Surgery of acute myocardial infarction-derived complications
* Other emergent cardiac surgeries (acute aortic dissection, heart injuries).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing heart surgery in our hospital from 2009 to June 2020. Patients were categorized in blood-transfusion non-acceptors (exposed cohort) and blood-transfusion acceptors (control cohort)
Sampling Method: Non-Probability Sample
Enrollment: 1911 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Change on Hemoglobin values from preoperative to end-of-surgery levels | End-of-surgery
  Changes on Hemoglobin values in percentage from preoperative level to the end of the surgery level

SECONDARY OUTCOMES:
Rate of operative mortality | At discharge or within the first 30 postoperative days
  Any death occurring i) within the first 30 postoperative days in or out of the hospital, and ii) after 30 days during the same hospitalization subsequent to the operation.
Intraoperative fluid balance | End of surgery
  Resting the fluid outputs to inputs
Hemoglobin at discharge | At discharge, an average of 10 days
  Hemoglobin level at discharge
Rate of postoperative morbidity | At discharge, an average of 10 days
  Postoperative complications: hemodynamic, respiratory, renal, neurological, infective complications

CONTACTS AND LOCATIONS:
Overall Officials: Elena Roselló-Díez, MD, PhD, Principal Investigator — Cardiac surgeon
Locations (1):
- Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Undecided